CLINICAL TRIAL: NCT06461728
Title: Minimal Instrumentation With Intracanal Heating ad Activation of Sodium Hypochlorite for
Brief Title: Minimal Instrumentation With Intracanal Heating and Activation of Sodium Hypochlorite for the Management of Teeth With Periapical Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USJ-2023-266
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Heating and Activation of Sodium Hypochlorite

STUDY DESIGN:
Intervention Model Description: Thirty-two single rooted teeth (N=32) with pulp necrosis and asymptomatic apical periodontitis
Who Masked: Participant
Masking Description: All patients will be recruited at the postgraduate Endodontics Clinic of the faculty of dentistry at Saint Joseph University. They will be given a patient health survey form and the ones who meet the inclusion criteria will take part of the study after a written informed consent form is obtained. All patients will be informed about the objectives, methods and follow-up by the same operator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator): Each canal will be prepared using Reciproc Blue nickel titanium file 25/08 and sonic activation of NaOCl
  Interventions: Device: a new prototye device that heat and activate sodium hyochlorite (Aseptico)
- conservative technique (Experimental): in the conservative technique, a size 10 FlexoFile will be introduced ,a glide path will be established using the size 10 FlexoFile to the WL, than Proglider 16.02 to the foramen.
  than heating and activation of NaOCl will be done with a prototype needle
  Interventions: Device: a new prototye device that heat and activate sodium hyochlorite (Aseptico)

INTERVENTIONS:
Device: a new prototye device that heat and activate sodium hyochlorite (Aseptico) — endoactivator : it is a sonic activator device
  Other Names: Endoactivator (in the conventional group ) -Dentsply

SUMMARY:
this study is the first to demonstrate the efficacy of minimally invasive root canal treatment combined with intracanal heating and activation of NaOCl using a prototype needle on the healing of asymptomatic apical periodontitis of necrotic single rooted teeth. 32 teeth will be randomaly assigned into 2 groups :conventional and conservative technique .In the conventional group : each canal will be prepared using Reciproc Blue 25/08, approximetly 27 ml of NaOCl will be used , the canal will be activated using 20.02 taper tip of a sonic decive . This cyclel will be repeated 3 times and the obturation will be done using a single cone technique with AH plus resin-based sealer . In the second group a size 10 k file will be introduced to confirm patency and to record working length after filling the canal with NaOCl. A glide path will be established using the size 10 FlexoFile to the WL, than Proglider 16.02 to the foramen. After the glide path, the canal will be irrigated with 3 ml of 5, 25 % of NaOCL .The prototype needle tip will be placed in the canal to the length that is a little shorter than the length at binding point , in order to heat and activate the irrigant solution for 30 seconds.Step one is repeated 4 more times and a fresh solution of NaOCl is replaced every time. Canals will be dried using sterile paper points size 15 and the obturation will be performed for all teeth using the same technique as group 1 but with a standardized gutta percha point 2% tapered

DETAILED DESCRIPTION:
32 single rooted teeth with pulp necrosis and asymptomatic apical periodontitis as confirmed by negative response to cold tests and the absence of bleeding on entering the pulp chamber also radiographs will be included in this study and the periapical status will be decided in accord with the periapical Index (PAI).

The endodontic procedure will be performed under strict aseptic settings and a dental operation microscopea. After confirming the clinical and radiological diagnosis, the access cavity will be performed using sterile round diamond ,then a size 10 FlexoFile (Dentsply, Maillfer, Ballaigues, Switzerland) will be introduced to confirm patency and to record working length after filling the canal with sodium hypochlorite.

Then a size 15 Flexofile (Dentsply,Maillfer,Ballaigues,Switzerland)will be introduced into the canal , only root canals with an initial apical size equivalent to 15 k file will be selected and roots with larger foramina will be excludedThen the teeth will be randomly assigned into two experimental groups(n=16): conventional or conservative technique.

Group 1: conventional rotary instrumentation. Each canal will be prepared using Reciproc Blue nickel titanium file 25/08 (VDW, Munich, Germany) according to the manufacturer's instructions. . Continuous checking of the canal patency will be done using size 10 hand file followed by irrigation with 3 ml of 5.25% sodium hypochlorite at room temperature using irriflex endodontic irrigation needle (Produits Dentaires SA, Vevey, Switzerland) mounted on a 3ml syringe (Plastipak, Franklin Lakes, NJ, USA). Each time the instrument will be removed out of the canal and before using the next instrument. Approximately, 27 ml of NaOCl will be used until Reciproc Blue reaches WL. Once the instrumentation is done, the canal will be irrigated with 5 ml of 17% ethylenediaminetetraacetic acid (EDTA) keeping it in the canal for 3 minutes and then flushed with 5 ml of saline.

In the end, the canal will be filled with 5.25% NaOCl at room temperature and and activated using the size 20 .02 taper tip of a sonic device (EndoActivator, Dentsply Tulsa Dental Specialties, Tulsa, OK, USA) at 10,000 cycles/min and the activator tip will be placed within 2 mm of the working length.

This cycle will be repeated three times and the canal will be rinsed with 3 ml of 5.25% NaOCl at room temperature after each cycle.

After the completion of the endodontic procedures, gauging of the apex will be done. The canals will be dried using sterile paper points size 25 (Maillfer,Ballaigues,Switzerland).

The obturation will be done using a single cone technique: AH plus resin-based sealer (Dentsply,DeTrey,Konstanz,Germany) will be mixed as per the manufacturer's instructions and applied to the root canal walls using a lentulo spiral also, the apical third of the gutta-percha size 25 (Maillfer,Baillaigues,Switzerland) will be coated with sealer and gently inserted into the canal to the working length. Excess of gutta-percha will be cut at the CEJ with a heat plugger (Fast-Pack pro-obturation system) and the coronal part of the gutta-percha will be condensed with gentle pressure using an endodontic plugger (Heat carrier Dentsply, Maillfer,Ballaigues,Switzerland).

Group 2: in the conservative technique, a size 10 FlexoFile (Dentsply,Maillfer,Ballaigues,Switzerland) will be introduced to confirm patency and to record working length after filling the canal with NaOCl. A glide path will be established using the size 10 FlexoFile to the WL, than Proglider 16.02 to the foramen. After the glide path, the canal will be irrigated with 3 ml of 5, 25 % of NaOCL at room temperature using irriflex endodontic needle (Produits Dentaires SA, Vevey, Switzerland) mounted on a 3ml syringe (Plastipak, Franklin Lakes, NJ, USA) .NaOCL is left in the canal and access cavity .The prototype needle tip will be placed in the canal to the length that is a little shorter than the length at binding point , in order to heat and activate the irrigant solution for 30 seconds . The tip will be moved with small (few mm) in-and out movement Than NaOCl will be aspirated from the canal and the access cavity than the canal will be filled with 17% EDTA, keeping it in the canal for 3 minutes followed by saline. Saline is aspirated. Step one is repeated 4 more times and a fresh solution of NaOCl is replaced every time. Canals will be dried using sterile paper points size 15 (Maillfer,Ballaigues,Switzerland) and the obturation will be performed for all teeth using the same technique as group 1 but with a standardized gutta percha point 2% tapered (Dentsply,Maillfer,Ballaigues,Switzerland) .

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients without any known allergic reactions or systemic diseases.
* Single rooted teeth.
* Fully formed roots.
* The ability to place #15 hand file to working length (WL).
* Absence of canal calcifications.
* Absence of root fracture.
* Absence of resorption.
* Teeth with pre-operative periapical radiolucency and PAI score ≥ 3 according to the classification of Ørstavik et al. 1986(20).
* Estimated WL 20-23mm.

Exclusion Criteria:

* Roots with broken or immature open apices.
* Roots presenting resorption.
* Patients younger than 18 years old.
* Pregnant patients.
* Teeth with previous root canal treatment.
* Teeth with calcified canals.
* Teeth with two canals or any other anatomic variations.
* Root length less than 16 mm.
* Patients with chronic generalized periodontitis.
* Teeth with caries affecting the roots.
* Abnormal mobility of the tooth.
* Extensively restored and prepared teeth.
* Open apices.
* Previously root canal therapy.
* Root cracks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
efficiency of minimal instrument combined with intracanal heating and activation of NaOCl | 3 , 6 and 9 months follow up
  evaluation of the clinical and radiographic healing of minimally invasive root canal treatment performed with minimal instrumentation combined with intra-canal heating and activation of NaOCl using a prototype needle on necrotic single rooted tooth with apical periodontitis compared to conventional root canal treatment with sonic activation by comparing the change of the area of the lesion

SECONDARY OUTCOMES:
To evaluate the speed of repair of healing periapical lesions | 3,6 and 9 months follow up
  To evaluate the speed of repair of healing periapical lesions, using the following formulas:
  Absolute speed of shrinkage (mm2/day) = ((initial detected area-final area))/(duration of treatment) Relative speed of shrinkage (per day)= ((initial detected area-final area) x 100)/(initial detected area x duration of the treatment )

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Any data will be shared with other researches if it is required or will help conducing further studies
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: the data are available at any time